CLINICAL TRIAL: NCT03098719
Title: GISMO - Geographical Information Support for Healthy Mobility
Acronym: GISMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Collaborators: University of Salzburg (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Professor of Medicine, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GISMO-1
Record Dates: First submitted 2017-03-18; First posted 2017-04-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Active Mobility
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Active Mobility — see detailed discription
  Arms: Intervention

SUMMARY:
GISMO combines spatial information with findings on the health effects of sustainable, active forms of mobility in the work environment in order to derive evidence-based decision-making bases for a health-promoting, operational mobility management. Existing approaches - with regard to spatial information systems, decision-support systems and health effects of active mobility - are considered and supplemented by our developments and investigations. Achieved non-personal results are provided through standardized web interfaces, ensuring integration into existing and prospective tools of an innovative and health-promoting mobility management.

DETAILED DESCRIPTION:
The World Health Organization recommends a minimum of 150 minutes per week of moderate activity as a minimum for a healthy daily routine. The average employee in Austria works on 5 days a week and covers the distance from his place of residence to his place of work twice. This distance can be actively traveled (e.g., bicycle) or passively (e.g., car).

Due to a moderate physical activity (intensity 4-6 METs, corresponding to 4-6 times resting energy conversion) of 15 minutes in one direction, only the active minimum requirement for everyday activity would be achieved by active mobility to and from the workplace.

Design:

2: 1 randomized controlled trial (intervention group: control group)

Activities:

Motivation of the employees by health care professionals of a sample company (Salzburger Landeskrankenanstalten AG, SALK) to use the public transport as well as the bicycle or footpath on the way from and to the workplace.

Intervention A: Change from car to bicycle for at least 50% of the routes, n = 20-25 Employees who have previously traveled exclusively by car and are living within a radius of ≤10 kilometers from the workplace are motivated by the GVPs to switch to a bicycle. In the case of appropriate proximity, employees can travel the entire path without motorized mobility. The greatest health benefit is to be expected by largely dispensing with motorized mobility at work. In the case of bad weather, cold or similar obstacles, a public transport or car can be used occasionally and exceptionally.

Intervention B: Exit from public transport one or more stations earlier or enter one or more station later, n = 20-25 By extending the path to and from a stop, which is to be actively pursued, a health effect is expected. In the context of this intervention, the availability of time tickets will provide incentives for switching from car to public transport. In addition, the employees are motivated to use the next stop in order to extend the active distance. Access routes can also be covered on foot.

Control group: Maintaining the mobility as before n = 20-25

Method:

Before and after the intervention phase of 1 year (to take into account seasonal effects or fluctuations), parameters relevant to health are collected. Finally, the results of the initial examination are compared with those of the final examination in order to examine the effects of healthy mobility on the workplace on cardiovascular risk profile, everyday activity, physical performance, quality of life, mobility behavior, body composition.

The aim of this project is to generate data on the health effects of a healthy mobility.

ELIGIBILITY:
Inclusion Criteria:

* employees of SALK (possibly also employees of other companies), age 18-70 voluntary participation in the study, consent in German language, desire to change the currently prevailing passive mobility behavior.

Exclusion Criteria:

* physical or psychological condition that makes the participation and completion of the study unlikely. i.e.:

  * Participation in further clinical trials at the same time, or at least four weeks time
  * Pregnancy or lactation
  * Well-known diseases of the movement apparatus, which could influence healthy mobility
  * Subjects with known endogenous or reactive depression or other psychiatric disorders such as panic disorder, schizophrenia, organic mental disorder, delirious, psychotic, phobic, or other psychiatric disorder in the last five years prior to study inclusion
  * Subjects with osteoporosis requiring treatment
  * Severe general disease (e.g., neoplasia, tuberculosis, heart failure)
  * Subjects with chronic infections
  * subjects with alcohol or drug abuse or dependency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness, i.e. metaboloic equivalents (METs) | 1 year
  Ergometry

SECONDARY OUTCOMES:
Cardiovascular Risk | 1 year
  Heart Score of the European Society of Cardiology

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No